CLINICAL TRIAL: NCT03256357
Title: Effectiveness of Intensive Upper Limb Training Combining Constraint-Induced Movement Therapy and Action Observation Training in Children With Unilateral Cerebral Palsy
Brief Title: Constraint-Induced Movement Therapy and Action Observation Training in Children With Unilateral Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Collaborators: ETH Zurich (Switzerland) (Other); University of Pisa (Other)
Responsible Party: Principal Investigator, Klingels Katrijn, Principal Investigator, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CIMT and AOT in unilateral CP
Record Dates: First submitted 2017-07-14; First posted 2017-08-22 (Actual); Last update posted 2019-10-28 (Actual); Status verified 2019-10

CONDITIONS: Cerebral Palsy
Keywords: unilateral cerebral palsy; upper limb rehabilitation
MeSH Terms: conditions — Cerebral Palsy | interventions — Constraint Induced Movement Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- CIMT + AOT (Active Comparator): In a 2-week day camp model children receive constraint-induced movement therapy for six hours a day, for 9 out of 11 consecutive days. All children wear a tailor made hand splint on the unaffected upper limb for 6 hours per day while performing unimanual exercises individually or in a group based on shaping and repetitive practice.
  Action observation training consists of 15 sessions of 1 hour. Children watch video sequences showing goal-directed actions and subsequently execute the observed actions with the affected upper limb.
  Interventions: Behavioral: Constraint-induced movement therapy; Behavioral: Action observation training
- CIMT + POT (Placebo Comparator): In a 2-week day camp model children receive constraint- induced movement therapy for six hours a day, for 9 out of 11 consecutive days. All children wear a tailor made hand splint on the unaffected upper limb for 6 hours per day while performing unimanual exercises individually or in a group based on shaping and repetitive practice.
  Placebo observation training consists of 15 sessions of 1 hour.This group performs the same actions after watching computer games without biological movements.
  Interventions: Behavioral: Constraint-induced movement therapy; Behavioral: Placebo observation training

INTERVENTIONS:
Behavioral: Constraint-induced movement therapy — In a 2-week day camp model children receive constraint- induced movement therapy for six hours a day, for 9 out of 11 consecutive days. All children wear a tailor made hand splint on the unaffected upper limb for 6 hours per day while performing unimanual exercises individually or in a group based on shaping and repetitive practice.
Behavioral: Action observation training — Action observation training consists of 15 sessions of 1 hour. Children watch 3 minute video clips of unimanual goal-directed actions followed by 3 minutes of execution of the actions.
  Arms: CIMT + AOT
Behavioral: Placebo observation training — Placebo observation training consists of 15 sessions of 1 hour. Children perform the same actions as the AOT training after watching computer games without biological movements.
  Arms: CIMT + POT

SUMMARY:
A randomized, controlled, and evaluator-blinded trail will be carried out comparing CIMT with or without AOT on sensorimotor outcome in children with unilateral CP aged 5 to 12 years. Additionally the potential role of neurological factors, including the anatomical characterization of the brain lesion, structural/functional connectivity and cortical reorganization, on treatment response will be investigated.

DETAILED DESCRIPTION:
Background: Problems in upper limb (UL) function in children with unilateral cerebral palsy (UCP) are traditionally trained with motor execution treatment models, such as Constraint Induced Movement Therapy (CIMT). However new approaches based on a neurophysiological model such as action observation training (AOT) may provide new opportunities for enhanced motor learning.

Aim: The aim of study is to investigate the effects of an intensive treatment model consisting of CIMT and AOT compared to CIMT alone on UL function in children with UCP. Additionally the potential role of neurological factors (including the anatomical characterization of the brain lesion, structural/functional connectivity and cortical reorganization) on treatment response will be analysed.

Methods/Design: A randomized, controlled, evaluator-blinded trial (RCT) will be conducted in 40 children between 5 and 12 years of age. Before randomization, children are stratified according to their House Functional Classification Scale, age and type of cortical reorganization. The Intervention is accomplished during a 2-week day camp in which the children receive intensive therapy for six hours a day on 9 out of 11 consecutive days (54 h) including AOT or placebo observation training (POT) (15h). During the AOT the children in the experimental group watch video sequences showing goal-directed actions and subsequently execute the observed actions with the affected UL. Children in the POT group perform the same actions after watching computer games without biological movements.

Outcome assessments include qualitative and quantitative measures of UL sensorimotor function across the International Classification of Functioning, Disability and Health (ICF). The primary outcome measure is the Assisting Hand Assessment (AHA). The medical imaging protocol includes structural Magnetic Resonance Imaging (MRI), Diffusion Kurtosis Imaging (DKI), resting state functional MRI (rs-fMRI) and Transcranial magnetic stimulation (TMS). The timeline for the assessment is T0 (1-1.5 month before the camp onset), T1 (before the intervention), T2 (after the intervention) and T3 (6 months after the intervention). Linear mixed models will be used to study time effects of the interventions and the interaction with neurological variables as covariates.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of unilateral CP
* aged 5-12 years
* sufficient cooperation to comprehend and complete the test procedure
* minimal ability to actively grasp and stabilize an object

Exclusion Criteria:

* upper limb surgery two years prior to enrollment
* botulinum toxin A injections six months prior to enrollment

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Change in Assisting Hand Assessment (AHA) | baseline, pre and post intervention (within one week), 6 months follow-up
  The AHA, a Rasch-based performance scale, measures how effectively the affected hand is spontaneously used during performance of bimanual tasks.

SECONDARY OUTCOMES:
Change in Melbourne Assessment of Unilateral Upper Limb Function | baseline, pre and post intervention (within one week), 6 months follow-up
  The Melbourne Assessment evaluates quality of movement in 16 functional unimanual tasks.
Change in Jebsen-Taylor Hand Function Test | baseline, pre and post intervention (within one week), 6 months follow-up
  The Jebsen-Taylor hand function test measures manual dexterity in six unimanual tasks, by means of movement time expressed in seconds for both hands.
Change in Tyneside Pegboard test | pre and post intervention (within one week), 6 months follow-up
  The Tyneside pegboard test is an adapted 9-hole pegboard test and assesses unimanual and bimanual dexterity.
Change in passive range of motion (PROM) | baseline, pre and post intervention (within one week), 6 months follow-up
  PROM of shoulder flexion, abduction, external and internal rotation, elbow extension, forearm supination and wrist extension is measured using a universal goniometer.
Change in muscle tone | baseline, pre and post intervention (within one week), 6 months follow-up
  Muscle tone is evaluated in 11 muscle groups using the Modified Ashworth Scale (MAS), ranging from 0 to 4.
Change in muscle strength | baseline, pre and post intervention (within one week), 6 months follow-up
  Muscle strength is evaluated in nine muscle groups using manual muscle testing (MMT), ranging from 0 to 5.
Change in grip strength | baseline, pre and post intervention (within one week), 6 months follow-up
  Grip strength is assessed with a Jamar dynamometer®. The average of three consecutive maximum contractions is recorded for both hands.
Change in muscle fatigability | baseline, pre and post intervention (within one week), 6 months follow-up
  Muscle fatigability during an isometric grip strength task is assessed based on a 30 second sustained contraction with E-link software.
Change in Abilhand-Kids questionnaire | baseline, pre and post intervention (within one week), 6 months follow-up
  The Abilhand- Kids questionnaire is a Rasch-based inventory of 21 mostly bimanual activities that the parents are asked to judge as: 0 (impossible), 1 (difficult), and 2 (easy), irrespective of the limb(s) actually used to do the activity.
Change in Children's Hand-use Experience Questionnaire (CHEQ) | baseline, pre and post intervention (within one week), 6 months follow-up
  CHEQ is a questionnaire to evaluate the experience of children and adolescents in using the affected hand in activities where usually two hands are needed.
Change in Upper limb Three-dimensional movement analysis (3DMA) | pre and post intervention (within one week), 6 months follow-up
  This quantitative assessment comprises upper limb kinematics during functionally relevant aiming and grasping tasks.
Change in Assessment of Life Habits for children (LIFE-H Kids) | pre intervention (within one week), 6 months follow-up
  LIFE-H Kids assesses the quality of social participation of children with disabilities by estimating how a client accomplishes activities of daily living and social roles
Change in Cerebral Palsy Quality of Life Questionnaire (CP-QOL) | pre intervention (within one week), 6 months follow-up
  CP-QOL is a parent report that assesses the wellbeing across various domains of life in children with cerebral palsy.

OTHER OUTCOMES:
Structural Magnetic Resonance Imaging (MRI) | baseline
  Structural images are acquired using three-dimensional fluid-attenuated inversion recovery (3D FLAIR) with following parameters: 321 sagittal slices, slice thickness 1.2, slice gap 0.6, repetition time=4800 ms, echo time=353 ms, field of view=250 x 250 mm², 1.1 x 1.1 x 0.56 mm³ voxel size, acq time = 5'02". Brain lesions will be first classified according to the timing of the lesion and the predominant pattern of damage as described by Kragelöh-mann (2007): cortical malformations (first and second trimester of pregnancy), periventricular white matter (PWM) lesions (from late second till early third trimester) and cortical and deep greymatter (CDGM) lesions (around term age) and acquired brain lesions (between 28 days 3 years postnatally). Second, a more detailed evaluation of the brain lesion (i.e. location and extent) will be performed using the semi-quantitative MRI (sqMRI) scale developed by Fiori et al. (2014).
Resting state functional Magnetic Resonance Imaging (rsfMRI) | baseline
  rsfMRI images are acquired using a T2*-weighted gradient-echo planar imaging (GE-EPI) sequence with the following parameters: TR = 1700 ms; TE = 30 ms; matrix size = 64x64; FOV = 230 mm; flip angle = 90º; slice thickness = 4 mm; no gap; axial slices = 30; number of functional volumes = 250; acquisition time = 7 min. rsfMRI will be pre-processed with Statistical Parametric Mapping version 12 (SPM12) software. Functional connectivity analysis will be computed with the CONN toolbox v17b.
Diffusion weighted imaging | baseline
  Diffusion weighted images will be acquired using a single shot spin echo sequence with the following parameters: slice thickness = 2.5 mm, TR = 8700 ms, TE = 116 ms, number of diffusion directions = 150, number of sagittal slices = 58, voxel size = 2.5 x 2.5 x 2.5 mm³, acq time = 18'. Implemented b values are 700, 1000, and 2800 s/mm², applied in 25, 40, and 75 uniformly distributed directions, respectively. In addition, 11 non-diffusion weighted images are obtained. Diffusion data will be pre-processed and analyzed in ExploreDTI toolbox, version 4.8.6. Diffusion metrics, such as fractional anisotropy and mean diffusivity of white matter tracts of interest (i.e. corpus callosum, corticospinal tract, superior thalamic radiations, medial lemniscus) will be calculated for both hemispheres.
Transcranial Magnetic Stimulation (TMS) | baseline
  TMS was performed using a MagStim 200 Stimulator (Magstim Ltd, Whitland, Wales, UK) equipped with a focal 70mm figure-eight coil and a Bagnoli electromyography (EMG) system with two single differential surface electrodes (Delsys Inc, Natick, MA, USA). A Micro1401-3 acquisition unit and Spike software version 4.11 (Cambridge Electronic Design Limited, Cambridge, UK) were used to synchronize the TMS stimuli and the EMG data acquisition. Motor Evoked Potentials (MEPs) were bilaterally recorded, using single differential surface EMG electrodes attached on the muscles adductor pollicis brevis of both hands.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Simon-Martinez, Principal Investigator — KU Leuven; Hilde Feys, Prof, Study Director — KU Leuven
Locations (1):
- KU Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Simon-Martinez C, Mailleux L, Hoskens J, Ortibus E, Jaspers E, Wenderoth N, Sgandurra G, Cioni G, Molenaers G, Klingels K, Feys H. Randomized controlled trial combining constraint-induced movement therapy and action-observation training in unilateral cerebral palsy: clinical effects and influencing factors of treatment response. Ther Adv Neurol Disord. 2020 Jan 6;13:1756286419898065. doi: 10.1177/1756286419898065. eCollection 2020. PMID 32031542
- [Derived] Simon-Martinez C, Mailleux L, Ortibus E, Fehrenbach A, Sgandurra G, Cioni G, Desloovere K, Wenderoth N, Demaerel P, Sunaert S, Molenaers G, Feys H, Klingels K. Combining constraint-induced movement therapy and action-observation training in children with unilateral cerebral palsy: a randomized controlled trial. BMC Pediatr. 2018 Jul 31;18(1):250. doi: 10.1186/s12887-018-1228-2. PMID 30064396